CLINICAL TRIAL: NCT06844123
Title: Graft Robot-Assisted Corneal Enhancement
Brief Title: Microsurgical Robot-assisted Corneal Transplant
Acronym: GRACE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PS25009*
Record Dates: First submitted 2025-02-06; First posted 2025-02-25 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Corneal Dystrophy
MeSH Terms: conditions — Corneal Dystrophies, Hereditary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Robot-assisted keratoplasty group (Experimental): patients undergoing robot-assisted corneal transplantation
  Interventions: Procedure: Robot-assisted keratoplasty

INTERVENTIONS:
Procedure: Robot-assisted keratoplasty — Feasibility pilot interventional study. Monocentric, one arm. Microsurgical robot will be used to perform penetrating keratoplasty. During the procedure, the corneal sutures will be performed using symani surgical system, that is a microsurgical robot controlled by a surgeon

SUMMARY:
Full-thickness corneal grafting (transfixing keratoplasty) is a tissue graft described at the beginning of the 20th century, which has remained technically unchanged for several decades. Around 900 transfixing keratoplasties are performed every year in France. This microsurgical procedure is intended for patients with severe corneal pathology that seriously impairs visual function, and for whom no therapeutic alternative - optical devices, medication or other surgical procedure - exists.

The initial anatomical outcome of surgery depends on the accurate execution of the corneal sutures. Very recently, a robot with microsurgical capabilities was developed by the MMI company (Symani® surgical system, now available from the Reims University Hospital). This robot is equipped with forceps and a needle holder capable of handling fragile tissues and microsurgical needles with an amplitude of movement greater than that of the human hand. It is operated by a surgeon via a wireless controller and foot pedal. It could thus be used to perform the usual sutures of a transfixing keratoplasty.

To our knowledge, no study to date has evaluated the contribution of a microsurgical robot to transfixing keratoplasty in humans. The Symani® microsurgical robot recently received CE marking for microsurgery. The investigators were able to carry out a series of ex vivo keratoplasties using the robot to suture non-conforming human corneas (destined for destruction), thus proving the feasibility of the procedure.

On the basis of this proof of concept, our project aims to evaluate the performance of robot-assisted transfixing keratoplasty in patients requiring corneal transplantation. Robotic assistance for human eye surgery, particularly corneal transplants, has never been evaluated. The use of a robot to perform corneal sutures during transfixing keratoplasty could equal or even surpass the performance of this crucial surgical step, which is conventionally performed manually. Ultimately, visual results could be equivalent or even better than those obtained after conventional surgery. At the same time, the use of the robot will be evaluated in terms of surgical cost, in order to obtain a quantified financial evaluation of robot-assisted keratoplasty.

DETAILED DESCRIPTION:
Context Transfixing keratoplasty was developed in the early 20th century. The aim is to replace the entire central cornea with a corneal allograft. This microsurgical procedure is performed with the aid of an operating microscope, and under general anesthetic to ensure optimal control of the absence of movement and arteriovenous pressure throughout the procedure.

Suturing is therefore an essential part of transfixing keratoplasty. They determine the congruence of the tissue edges and the distribution of tension applied to the sutures, thus modulating the curvature (astigmatism) of the graft. This curvature will determine the optical properties of the eye, and hence its acuity and the patient's visual recovery. A topical immunomodulatory local treatment (corticosteroids and/or ciclosporin eye drops) is administered for several years; no systemic treatment is used. Sutures are usually removed 6 months to 1 year after surgery. Current indications are major declines in visual acuity - generally below 4/10 with the best possible correction - associated with i) severe keratoconus, the most frequent indication, ii) failed anterior grafts, iii) full-thickness central corneal scars, and iv) hereditary stromal dystrophies.

Robot-assisted surgery has developed considerably over the last twenty years, with procedures now routinely performed in macro- and endoscopic surgery (mainly urology, obstetrics and visceral surgery). Very recently, engineering advances in precision motion control and mechanical miniaturization have enabled the development of robots dedicated to microsurgery. The Symani® Surgical System (Medical MicroInstrument, Pisa, Italy) has been used and evaluated in animals and humans over the past two years for vessel and nerve microsurgery. The Symani® robot is equipped with forceps and a needle holder capable of handling fragile tissue, as well as microsurgical needles and wires (8/0 to 12/0). The Symani® robot has recently been CE-marked for microsurgery [appendix 1]. To date, there is only one study - ex vivo and in animals - on the feasibility of its use in ocular surgery. On the basis of the robot's capabilities and its CE mark, the investigators have carried out preliminary experiments, enabling us to envisage robot-assisted keratoplasty in humans.

On the basis of our preliminary results, the investigators hypothesize that it is possible to use the Symani® robot's assistance to perform the major surgical stage of transfixing keratoplasty, i.e. the sutures between the graft and the recipient cornea, in humans.

Objectives :

* Main:

  1. Evaluate the feasibility, and intraoperative intercurrent events of robotic assistance during transfixing keratoplasty,
  2. Identify possible early and late postoperative intercurrent events/adverse events related to robot use.
* Secondary :

  i) Evaluate the impact of robotic assistance during transfixing keratoplasty on postoperative corneal anatomical outcome (graft curvature).

ii) Assess the impact of robotic assistance on refraction and visual outcome in the medium term: 3 months iii) Evaluate the mean degree of astigmatism post robotic-assisted grafting, so as to be able to calculate the number of subjects required for a subsequent study of the superiority of robotic-assisted surgery over usual conventional surgery.

iiii) Evaluate the additional cost of robotic-assisted surgery. iv) Evaluate the quality of life before and 3 months after the intervention Type of study: pilot feasibility study, monocentric, interventional. Population: Ten consecutive adult patients requiring transfixing keratoplasty who agreed to participate by signing an informed consent form.

Investigation plan : The study will be offered to patients scheduled for penetrating keratoplasty. Clinical follow-up will be conducted at Day 1, Day 7, Day 30. Final clinical and paraclinical check-up at Day 90 and end of participation.

ELIGIBILITY:
inclusion criteria :

* Patients of legal age seen in a specialized ophthalmology consultation at the Reims University Hospital, and requiring transfixing keratoplasty.
* Affiliated to a social security scheme
* Agreeing to take part in the study (information and signature of consent form).

exclusion criteria :

* Patients protected by law
* Patients with an ocular pathology other than their corneal pathology.
* Mentally incapable of adhering to the principles of the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Descriptive analysis of unusual events intra- and postoperatively | Day O (intraoperative) to Day 7
  Number and percentage of unusual events
Descriptive analysis of unusual events | Day 7 to Day 90
  Number and percentage of unusual events

SECONDARY OUTCOMES:
Postoperative corneal anatomical result | Day 90
  Anterior topographic will be performed and compare central astigmatism
Visual acuity with correction | Day 90
  The mean diopters
Visual acuity without correction | Day 90
  The mean diopters
Corneal topographic regularity | Day 90
  Corneal topographic regularity measured by surface regularity index (SRI)
Corneal topographic regularity | Day 90
  Corneal topographic regularity measured by surface asymmetry index (SAI)
Subjective refraction | Day 90
  Measurement of spherical equivalent (SE)
Subjective refraction | Day 90
  Measurement of refractive astigmatism (CYL)
Analysis of surgical costs | Month 6
  cost of graft and materials used
National Eye Institute Visual Function Questionnaire | Day 90
  Quality of life - National Eye Institute Visual Function Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France